CLINICAL TRIAL: NCT06317402
Title: Evaluate the Prevalence of Undernutrition in Adult Patients Hospitalized on a Given Day at the Pitié-Salpêtrière Hospital (PSL) According to HAS Criteria in 2019 (if Age <70 Years) and 2021 (if Age ≥ 70 Years)
Brief Title: Epidemiology and Management of Malnutrition of Patients Hospitalized at the Pitié-Salpêtrière Hospital: a One-day Survey Combined With Focus Groups (Mixed Methods)
Acronym: EPIDENUT_PSL
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP240133
Record Dates: First submitted 2024-03-12; First posted 2024-03-19 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Malnutrition
Keywords: malnutrition
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- patient: Adult patients hospitalized at Pitié Salpêtrière in conventional hospitalization wards
  Interventions: Other: malnutrition questionary

INTERVENTIONS:
Other: malnutrition questionary — At the patient's bed, using a questionnaire, evaluators take anthropometric measurements (weight, height, muscle strength) and collect biological data (albumin, pre-albumin, CRP, if available in the medical record) to establish nutritional status according to HAS criteria for undernutrition 2019-2021 and 2003-2007.

SUMMARY:
According to the literature, malnutrition affects between 30% and 50% of hospitalized patients. The most recent survey on the prevalence of malnutrition in hospitals in France dates back to 2003, and at the Pitié Salpêtrière Hospital to 2015. Malnutrition is a pathological process that can lead to complications for patients and prolong their length of stay.

Main objective: Evaluate the prevalence of malnutrition in adult patients hospitalized on a given day at Pitié-Salpêtrière Hospital (PSL) according to HAS ( High Authority for Health) criteria for 2019 (if age <70 years) and 2021 (if age ≥ 70 years).

DETAILED DESCRIPTION:
According to the literature, malnutrition affects between 30% and 50% of hospitalized patients. The most recent survey on the prevalence of malnutrition in hospitals in France dates back to 2003, and at the Pitié Salpêtrière Hospital to 2015. Malnutrition is a pathological process that can lead to complications for patients and prolong their length of stay.

Main objective: Evaluate the prevalence of malnutrition in adult patients hospitalized on a given day at Pitié-Salpêtrière Hospital (PSL) according to HAS (High Authority for Health) criteria for 2019 (if age <70 years) and 2021 (if age ≥ 70 years).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Hospitalized for at least 2 days in a Pitié Salpêtrière department of the 8 selected DMUs.
* Patient informed and not objecting to participation in the study.

Exclusion Criteria:

* Be hospitalized in a PRM, SMR, radiotherapy or adult psychiatry department
* Be hospitalized in an intensive care or resuscitation unit of the 8 selected DMU
* Be at the end of life, as determined by the referring clinician
* Have a communication barrier preventing the collection of declarative data
* Pregnancy in progress; 6. Patient under guardianship.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients hospitalized at Pitié Salpêtrière in conventional hospitalization wards (medical and surgical wards)
Sampling Method: Non-Probability Sample
Enrollment: 385 (Estimated)
Dates: Start 2024-05-15 (Actual); Primary Completion 2025-09-09 (Estimated); Study Completion 2025-09-09 (Estimated)

PRIMARY OUTCOMES:
Prevalence of undernutrition diagnosed according to HAS 2019 and 2021 criteria on a given day in hospitalized PSL patients. | 3 days
  The survey is conducted over 3 days due to : - The mobilization of medical and paramedical staff for the undernutrition screening phase is only possible over a limited period of time. - The patients to be assessed will be drawn at random from a list provided by the Admissions department ; the draw will then be carried out by the Public Health department (excluding the ORIGYNE DMU, the PRM and respiratory and neurorespiratory SSR departments, and the radiotherapy department (few hospitalizations lasting more than 24-48 hours)). In addition, it is important to specify that, if at the end of phase 1 of the survey, the auditor (dietician and/or doctor) finds that a patient is undernourished, the auditor will inform the department's referring doctor within 24 hours. The resulting treatment will be carried out by the referring dietician on the basis of a medical prescription.

SECONDARY OUTCOMES:
Compare the prevalence and the severity of undernutrition in hospitalized PSL patients according to the HAS criteria of 2019 (if age <70 years) and 2021 (if age ≥ 70 years) versus those of 2003 (if age <70 years) and 2007 (if age ≥ 70 years). | 6 months
  Phase 1 : HAS malnutrition criteria 2019-2021 and 2003-2007.
Evaluate the quality of nutritional management for malnourished patients hospitalized at PSL. Using PMSI coding, assess the value of activities associated with undernutrition in undernourished patients hospitalized at PSL. | 6 months
  Phase 2 : The quality of nutritional management of malnourished patients will be assessed using several judgment criteria extracted from patient records in Orbis, for the sub-group of patients hospitalized on the given day and diagnosed as malnourished during the 1st evaluation phase. Phase 3: Transmission of the list of NIP.IPP codes for patients diagnosed as undernourished to the DIM (Département d'Information Médicale) team for extraction of codes for diagnosis of undernutrition and procedures associated with its management.

CONTACTS AND LOCATIONS:
Overall Officials: Pauline Faucher, Dr, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Service de nutrition, Hôpital Pitié-Salpêtrière, Paris, France, France